CLINICAL TRIAL: NCT05809336
Title: Gut Microbial Metabolites Inosine Combined With PD-1/PD-L1 Inhibitor for Patients With Malignant Advanced Solid Tumors
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beijing inosine
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Inosine; camrelizumab; Injections; sintilimab; penpulimab; tislelizumab; pembrolizumab; toripalimab; atezolizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inosine group (Experimental): Participants will receive inosine + PD-1/PD-L1 inhibitor ± chemotherapy/targeting,every 2 or 3 weeks, until the subject's disease progresses, death, intolerable adverse events, the investigator determines that there is no benefit from continued treatment or other termination criteria are met (pregnancy, individual patient reasons or co-morbidities), the subject requests withdrawal from the study, withdrawal of informed consent, and loss of visit
  Interventions: Drug: Inosine 0.2g orally 3 times/day
- non-inosine group (Active Comparator): Participants will receive PD-1/PD-L1 inhibitor ± chemotherapy/targeting, every 2 or 3 weeks .until the subject's disease progresses, death, intolerable adverse events, the investigator determines that there is no benefit from continued treatment or other termination criteria are met (pregnancy, individual patient reasons or co-morbidities), the subject requests withdrawal from the study, withdrawal of informed consent, and loss of visit
  Interventions: Drug: PD-1/PD-L1 inhibitor ,chemotherapy/targeting

INTERVENTIONS:
Drug: Inosine 0.2g orally 3 times/day — inosine + PD-1/PD-L1 inhibitor ± chemotherapy/targeting,
  Other Names: Camrelizumab for injection; Sintilimab injection; Penpulimab injection; Tislelizumab injection; Pembrolizumab injection; Toripalimab; Atezolizumab; chemotherapy/targeting
  Arms: inosine group
Drug: PD-1/PD-L1 inhibitor ,chemotherapy/targeting — PD-1/PD-L1 inhibitor ± chemotherapy/targeting
  Other Names: Camrelizumab for injection; Sintilimab injection; Penpulimab injection; Tislelizumab injection; Pembrolizumab injection; Toripalimab; Atezolizumab; chemotherapy/targeting
  Arms: non-inosine group

SUMMARY:
We conducted a single-center, prospective randomized ,Parallel controls, open labels Clinical Studies,The study is about Gut Microbial Metabolites Inosine Combined With PD-1/PD-L1 Inhibitor for Patients with malignant Advanced Solid Tumors .One group was the inosine group , the other group was the non-inosine group.The treatment regimen of inosine group : inosine + PD-1/PD-L1 inhibitor ± chemotherapy/targeting, and the treatment regimen of non-inosine group : PD-1/PD-L1 inhibitor ± chemotherapy/targeting.The primary study endpoints were overall survival (OS) and progression-free survival PFS, and the secondary study endpoints were objective remission rate (ORR) and disease control rate (DCR) comparing the two groups.

DETAILED DESCRIPTION:
We conducted a single-center, prospective randomized ,Parallel controls, open labels Clinical Studies,,The study is about Gut Microbial Metabolites Inosine Combined With PD-1/PD-L1 Inhibitor for Patients with malignant Advanced Solid Tumors.One group was the inosine group , the other group was the non-inosine group. A total of 172 patients with advanced malignant solid tumors were collected from Capital Medical University Beijing Friendship Hospital, and randomly assigned to two groups according to 1:1, 86 patients in the inosine group and 86 patients in the non-inosine group. The regimen of inosine treatment group was: inosine + PD-1/PD-L1 inhibitor ± chemotherapy/targeting, and the treatment regimen of non-inosine treatment group was: PD-1/PD-L1 inhibitor ±chemotherapy/targeting,every 2 or 3 weeks protocol ,until the subject's disease progresses, death, intolerable adverse events, the investigator determines that there is no benefit from continued treatment or other termination criteria are met (pregnancy, individual patient reasons or co-morbidities), the subject requests withdrawal from the study, withdrawal of informed consent, and loss of visit.Anti-tumor efficacy is evaluated every 2/3 cycles (every 6 weeks) based on computed tomography (CT) or magnetic resonance imaging (MRI) results and their tumor markers, according to RECIST v1.1 criteria.

Inosine tablets were purchased from Tianjin Jinshi, dosage: 0.2g orally 3 times/day, PD-1/PD-L1 inhibitors, chemotherapy and targeted combination therapy regimens were developed by the investigators according to the NCCN guidelines and CSCO guidelines and the patient's condition and its staging.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed unresectable locally advanced, recurrent or metastatic solid tumors
2. Age 18 years old - 75 years old
3. ECOG score of ≤ 2
4. Time to end of palliative treatment for localized lesions (non-target lesions) was >3 weeks from randomization start time, At least one measurable lesion or assessable lesion according to RECIST v1.1
5. Can provide archived pathological tissues or fresh pathological tissues for PD-L1, MMR/MSI, TMB testing within 6 months from the signing of the informed consent for screening and can obtain the test results
6. Adequate organ and bone marrow function, defined as follows: 1) Blood count: absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 100 × 109/L, hemoglobin level (HGB) ≥ 9.0 g/dL. 2) Liver function: patients without liver metastases require: serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal ( ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN. patients with liver metastases required: TBIL ≤1.5×ULN; ALT and AST ≤5×ULN. 3) renal function: creatinine clearance (Ccr) ≥50mL/min (calculated using the Cockcroft/Gault formula): female: Ccr = (140-years-old) × body weight (kg) × 0.85; men: Ccr = (140-years-old) × body weight (kg) × 1.00. 4) Adequate coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5 × ULN
7. Expected survival time ≥ 12 weeks
8. Female subjects of childbearing age or male subjects whose sexual partners are women of childbearing age are required to use effective contraception throughout the treatment period and for 6 months after the treatment period
9. Sign the written informed consent

Exclusion Criteria:

1. Signs of active bleeding or perforation
2. History of intestinal obstruction or the following diseases: inflammatory bowel disease or extensive bowel resection, Crohn's disease, ulcerative colitis
3. Hepatic metastatic focal load of approximately 50% or more of the entire liver volume
4. Antibiotic was used within 2 weeks before study treatment
5. Received systemic antitumor therapy with herbs or immunomodulatory drugs (including thymidine, interferon, interleukin, etc.) within 2 weeks before the first dose.
6. immunosuppressive drugs was used within 4 weeks before study treatment, excluding topical glucocorticoids or physiologic doses of systemic glucocorticoids (i.e., no more than 10mg/day of prednisone or equivalent doses of other glucocorticoids) of nasal spray, inhalation, or other routes, or glucocorticoid for the prevention of contrast allergy
7. Interstitial lung disease requiring glucocorticoid therapy
8. Active, known or suspected autoimmune disease or history of the disease within the last 2 years (patients with vitiligo, psoriasis, alopecia or Grave's disease not requiring systemic treatment within the last 2 years, hypothyroidism requiring only thyroid hormone replacement therapy, and type I diabetes requiring only insulin replacement therapy may be enrolled)
9. Symptomatic congestive heart failure (New York Heart Association class -≥3) or symptomatic or poorly controlled arrhythmias
10. standard treatment could not uncontrollarterial hypertension (systolic blood pressure ≥ 160 or diastolic blood pressure ≥ 100).
11. Any arterial thromboembolic event, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, within 6 months prior to enrollment in treatment
12. History of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolism within 3 months prior to enrollment
13. Known active tuberculosis
14. Known history of case type immunodeficiency virus infection
15. Positive hepatitis B surface antigen and peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) titer test ≥ 1×104 copies/mL (or HBV-DNA quantification ≥ 2000 units/ml); active hepatitis C
16. History of other primary malignancies, except: malignancies in complete remission for at least 5 years prior to enrollment and requiring no other treatment during the study period; adequately treated non-melanoma skin cancer or malignant freckled nevus with no evidence of disease recurrence; adequately treated carcinoma in situ with no evidence of disease recurrence
17. Patients who, in the judgment of the investigator, are otherwise likely to interfere with the conduct of the clinical study, who may not be able to comply with the protocol or who are unable to cooperate, or who are a risk to the study This study was approved by the Clinical Investigation Ethics Committee of Beijing Friendship Hospital, Capital Medical University, and was conducted in accordance with the Declaration of Helsinki. All patients signed informed consent forms for data collection and study purposes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | 36 months
  Time from randomization grouping to death from any cause
progression-free survival (PFS) | 36 months
  Time from randomization grouping to the first recorded disease progression or death from any cause

SECONDARY OUTCOMES:
objective remission rate(ORR) [ Time Frame: Up to 36 months ] | 36 months
  Proportion of subjects with best overall efficacy assessed as CR and PR
disease control rate (DCR) | 36 months
  Proportion of subjects with best overall efficacy assessed as CR, PR and SD

CONTACTS AND LOCATIONS:
Locations (1):
- Qin li, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhao H, Zhang W, Lu Y, Dong Y, He Z, Zhen H, Li Q. Inosine enhances the efficacy of immune-checkpoint inhibitors in advanced solid tumors: A randomized, controlled, Phase 2 study. Cancer Med. 2024 Sep;13(17):e70143. doi: 10.1002/cam4.70143. PMID 39267574